CLINICAL TRIAL: NCT03669445
Title: Toward a Risk-adapted Strategy to Cure Myeloma : An Intensive Program With Lenalidomide, Ixazomib, and Dexamethasone Plus Daratumumab as Extended Induction and Consolidation Followed by Lenalidomide Maintenance in Newly Diagnosed Standard Risk Multiple Myeloma Patients Eligible for Autologous Stem Cell Transplant : a Phase II Study of the Intergroupe Francophone du Myélome (IFM)
Brief Title: Study Association of Lenalidomide, Ixazomib, Dexamethasone and Daratumumab in Newly Diagnosed Standard Risk Multiple Myeloma
Acronym: IFM2018-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/18/0212
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple myeloma; Daratumumab; Lenalidomide; Ixazomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- four drugs combination (Experimental): 21-day cycles induction, then 28-day cycles consolidation and maintenance with Lenalidomide, Ixazomib, and Dexamethasone Plus Daratumumab
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Ixazomib — 21-day cycles induction and 28-day cycles consolidation
Drug: Lenalidomide — 21-day cycles induction and 28-day cycles consolidation and 28-day cycles maintenance therapy
Drug: Dexamethasone — 21-day cycles induction and 28-day cycles consolidation
Drug: Daratumumab — 21-day cycles induction and 28-day cycles consolidation

SUMMARY:
The main objective of this study is to evaluate the minimal residual disease-negativity rate after administration of the combination of Lenalidomide, Ixazomib, Dexamethasone and Daratumumab as induction and consolidation therapy in an intensive program in newly diagnosed standard risk multiple myeloma patients.

For the induction therapy, each patient received 6 cycles of Lenalidomide, Ixazomib, Dexamethasone and Daratumumab, then peripheral blood stem cell harvest, intensification with autologous stem cell transplantation, consolidation therapy and maintenance.

DETAILED DESCRIPTION:
This is a phase II, multicenter, non-randomized, open-label study to evaluate the safety and efficacy of Lenalidomide, Ixazomib, Dexamethasone, and Daratumumab in patients with newly diagnosed multiple myeloma.

The patient population will consist of adult men and women ≤ 65 years, who have a confirmed diagnosis of standard risk multiple myeloma, who meet eligibility criteria.

Treatment periods will be defined as 21-day cycles for induction, and 28-day cycles for consolidation, and maintenance. Patients will be seen at regular treatment cycle intervals while they are participating in the study.

Patients will be assessed for disease response and progression according to the International Myeloma Working Group criteria at each cycle during induction and consolidation and every other cycle during maintenance.

Eastern Cooperative Oncology Group performance status, adverse events, laboratory values, and vital sign measurements will be collected and assessed to evaluate the safety of therapy throughout the study.

Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events. Patients will attend an End of Treatment visit after receiving their last dose of study drug and will continue to be followed for other follow-up assessments specified in the Schedule of events.

All patients will be followed for survival after progression.

ELIGIBILITY:
Inclusion Criteria:

* De novo symptomatic myeloma on the International Myeloma Working Group Diagnostic Criteria for the Diagnosis of Multiple Myeloma
* Measurable disease requiring systemic therapy defined by serum M-component ≥ 10g/l or urine M-component ≥ 200 mg/24h or involved free light level ≥ 100 mg/l
* Eastern Cooperative Oncology Group performance status 0, 1 or 2
* Eligible to high dose therapy

Exclusion Criteria:

* Previously treated with any systemic therapy for multiple myeloma
* Clinical signs of central nervous system involvement
* Renal insufficiency defined as estimated Glomerular Filtration Rate lower or equal to 40 ml/min/1.73 m2
* Hepatic impairment defined as aspartate transminase or alanine transaminase greater or equal to 3 x upper limit of normal, or Total bilirubin greater or equal to 3 x upper limit of normal
* Platelet count < 75,000 per µL
* Absolute neutrophil count ≤ 1,000 cells/mm3
* Evidence of current uncontrolled cardiovascular conditions
* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before first dose of study drug
* Grade 3 or higher peripheral neuropathy, or grade 2 with pain, on clinical examination during the screening period
* Known or suspected chronic obstructive pulmonary disease with a Forced Expiratory Volume in 1 second < 50% of predicted normal
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort within 14 days before initiation of the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
minimal residual disease-negativity rate | 22 months
  after completion of the consolidation therapy and before maintenance

SECONDARY OUTCOMES:
Adverse events | up to 54 Months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Response rates | 3 months, 5 months, 7 months, 13 months, 25 months
  Response rates according to the IMWG criteria after induction, high dose Melphalan, consolidation and maintenance therapy
Progression free survival | 54 months
Overall survival | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, Study Director — University Hospital, Toulouse
Locations (12):
- France (12):
  - CHU Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - University Hosptial Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided